CLINICAL TRIAL: NCT07254975
Title: An Observational Prospective Study of Anesthetic Sensitivity Assessed by Alpha Band Power and Its Association With Emergence Time From Sevoflurane General Anesthesia in Young Adults.
Acronym: ALPHA-SET
Status: Not yet recruiting | Type: Observational
Sponsor: University of Chile (Other)
Collaborators: Center for Advanced Clinical Research (CICA ) - University of Chile (Unknown)
Responsible Party: Sponsor
Other Study IDs: OAIC: 1526/25
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-10

CONDITIONS: Emergence From Anesthesia; EEG Power Spectra
Keywords: emergence from anesthesia; general anesthesia; sevoflurane; alpha power

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Young adults: Young adults (35-50 years) undergoing general anesthesia
  Interventions: Procedure: Intraoperative EEG Recording

INTERVENTIONS:
Procedure: Intraoperative EEG Recording — Patients will be monitored with a frontal EEG during general anesthesia using the BIS Monitor to calculate alpha power

SUMMARY:
The goal of this observational study is to determine the relationship between brain activity patterns and recovery time in adult patients (ages 35-50, ASA I-II) undergoing elective general anesthesia.

The main question it aims to answer is:

- Does a lower magnitude of intraoperative alpha wave power correlate with a longer time for patients to emerge from general anesthesia?

Participants will:

* Undergo a standardized general anesthesia (GA) protocol for elective surgery.
* Have their EEG activity recorded using a standard clinical BIS™ anesthetic depth monitor during the procedure.
* Have their time to awakening precisely measured after the cessation of anesthetic gases.

DETAILED DESCRIPTION:
General anesthesia (GA) is an essential technique in modern medicine, used to induce unconsciousness, analgesia, and immobility in patients during surgical procedures. Since no single drug can achieve all these conditions, a combination of agents acting on the central nervous system (CNS) is employed. These include GABAergic hypnotics, such as propofol and halogenated gases; opioids, such as remifentanil and fentanyl; and neuromuscular blocking agents, such as rocuronium. The co-administration of these drugs generates multiple interactions that allow anesthesia to be induced and maintained under predictable conditions, solidifying the concept of "balanced anesthesia." However, one of the major challenges in its management is the adequate titration of drugs according to the individual needs of each patient, in order to avoid both overdosing and underdosing, both of which pose potential risks to patient safety.

In this context, electroencephalography (EEG) has emerged as a key tool for monitoring anesthetic depth, providing real-time information on cerebral activity. The analysis of electroencephalographic patterns and spectrograms, particularly alpha wave power, has proven to be a useful indicator of the degree of decreased cerebral activity during general anesthesia. Furthermore, previous studies suggest that alpha wave power may correlate with anesthesia recovery time (Gutierrez et al., Anesthesia & Analgesia, 2021) and possibly with individual sensitivity to general anesthetics. However, this relationship has not yet been fully elucidated, as a systematic study confirming this correlation has not been conducted. Establishing a correlation between emergence time and alpha band power would allow us to determine individual sensitivity to the effects of general anesthetics.

General Objective:

To determine whether patients who are more sensitive to the effects of general anesthetics have a lower relative power in the alpha band and a longer emergence time from general anesthesia.

Specific Objectives:

1. - To quantify the relative alpha power in the electroencephalogram (EEG) spectrogram using an anesthetic depth monitor during the maintenance phase of general anesthesia in the study cohort.
2. - To precisely record the anesthetic emergence time, defined as the interval from the cessation of volatile anesthetic administration to the patient's recovery of consciousness (e.g., eye opening or response to verbal command).
3. - To statistically determine the correlation and magnitude of association between the quantified relative alpha power and the measured anesthetic emergence time.

Working Hypothesis Patients exhibiting greater cerebral sensitivity to general anesthetics, as indicated by a lower magnitude of relative alpha power during the maintenance phase, will experience a statistically significant prolongation of the anesthetic emergence time.

Methodology Materials and Methods: Subjects Following approval by the Ethics Committee of the Hospital Clínico Universidad de Chile, we will conduct an observational study on a cohort of patients undergoing general anesthesia. Given that only parameters obtained from a monitor and the time it takes for a patient to recover consciousness will be observed, an exemption from obtaining informed consent was approved by the ethics committee.

Study Protocol Patients will undergo conventional general anesthesia without major interventions. A BIS™ anesthetic depth monitor, which is routinely used in clinical practice, will be utilized to record anesthetic depth. The anesthesiologist will be requested to document the drugs used and to maintain general anesthesia, as is normally performed at our hospital, with sevoflurane at a standard dose of 0.8 to 0.9 MAC. Once the surgery is finished and anesthetic emergence begins, the minute the sevoflurane supply is stopped will be recorded. The moment consciousness is recovered, determined by eye opening and response to verbal or tactile stimuli (as is typically done in all general anesthetics), will be recorded.

In detail, a traditional general anesthetic at the Hospital Clínico de la Universidad de Chile consists of:

* Intravenous bolus administration of fentanyl at a dose of 3 mcg/kg.
* Subsequently, intravenous lidocaine administration at a bolus dose of 1 mg/kg, followed by the administration of an intravenous bolus of propofol at a dose of 2 mg/kg.
* Once the patient loses consciousness, the NMBA IV is administered at a dose of 0.6 mg/kg of rocuronium.
* The patient is then orotracheally intubated and connected to a mechanical ventilator.
* Anesthetic maintenance is achieved with sevoflurane and repeated doses of fentanyl and/or rocuronium as needed.
* Basic and necessary monitoring at all times consists of an electrocardiogram, pulse oximetry, capnography, intermittent non-invasive blood pressure, and anesthetic depth monitoring.
* For anesthetic emergence, the effect of neuromuscular blockers must be reversed, and sevoflurane is eliminated until the patient recovers consciousness.

As this is an observational study, the clinician responsible for the patient will administer the drugs they deem necessary and perform the relevant clinical measures; we will only record these actions.

Statistics A descriptive statistical analysis will be performed for each type of variable, expressing the results as percentages, medians, or means as appropriate. The records from the anesthetic depth monitor will be analyzed using MATLAB to determine the magnitude of the power in the alpha band. The sample size was calculated assuming that the alternative hypothesis (H1) for the linear correlation between alpha power and emergence time is r² = 0.4 ± 0.3, while the null hypothesis (H0) is r² = 0. Considering a statistical power of 90%, an alpha error of 0.05, a two-tailed analysis, and a possible loss of 20% of the data, it was determined that 70 patients are required (calculation performed with G*Power 3.1.9.4). Statistical analyses will be conducted using GraphPad Prism and R.

ELIGIBILITY:
Inclusion Criteria

* Elective surgery under general anesthesia
* Age 35-50 years
* ASA physical status I-II

Exclusion Criteria

* Neurological or psychiatric disorders
* Use of psychotropic drugs or opioids
* Altered consciousness
* BMI > 35 kg/m²
* Renal, cardiac, or hepatic dysfunction
* Emergency surgery
* Pregnancy
* Regional anesthesia

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Young adult patients undergoing an elective surgery at the Hospital Clínico, University of Chile, Santiago, Chile.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-11-24 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Anesthesia emergence time | 60 minutes
  Minutes from the end of the sevoflurane administration until eye opening to verbal stimulus

SECONDARY OUTCOMES:
Relative alpha power | 60 minutes
  Relative alpha power from the frontal EEG under general anesthesia
Absolute alpha power | 60 minutes
  Absolute alpha power from frontal EEG under general anesthesia
Extubation time | 60 minutes
  Time from the end of administration of sevoflurane until extubation
Fentanyl requirements | 1 day
  Total dose of fentanyl (mcg) requirement during general anesthesia
Propofol requirements | 1 day
  Total dose of propofol (mg) during general anesthesia
Sevoflurane requirement | 1 day
  Total dose of sevoflurane (mL) used during general anesthesia
Relative delta power | 1 day
  Relative delta power from frontal EEG under general anesthesia
Excitation and inhibitory EEG balance | 1 day
  Excitation/inhibition balance from frontal EEG under general anesthesia
Burst suppression time | 1 day
  Cumulative burst suppression time during general anesthesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gutierrez RG, Egana JI, Maldonado FA, Saez IA, Reyes FI, Soulat H, Purdon PL, Penna A. Association Between Lower Preoperative Cognition With Intraoperative Electroencephalographic Features Consistent With Deep States of Anesthesia in Older Patients: An Observational Cohort Study. Anesth Analg. 2021 Jul 1;133(1):205-214. doi: 10.1213/ANE.0000000000005262. PMID 33177327